CLINICAL TRIAL: NCT00945386
Title: The Effect of Continuous, Various Dosages of Furosemide Drip on Hearing as Measured by Acoustic Emission
Brief Title: The Effect of Continuous, Various Doses of Furosemide Drip on Hearing as Measured by Acoustic Emission
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Rabin Medical Center (Other)
Responsible Party: Dr. Elhanan Nahum, Rabin Medical Center
Other Study IDs: 005418
Record Dates: First submitted 2009-07-23; First posted 2009-07-24 (Estimated); Last update posted 2009-07-24 (Estimated); Status verified 2009-07

CONDITIONS: Hearing Status
Keywords: children; critically ill; furosemide; acoustic emission
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Pediatric patients, during their illness often treated with furosemide (Lasix) continuous drip, often, with dosages above 4-6mg/kg/day (the recommended dose).

This study will monitor hearing status of these children prior to their therapy with furosemide, during this therapy and after.

DETAILED DESCRIPTION:
This study will record hearing status, by acoustic emission, of critically ill children, treated with different dosages of furosemide drip.

Acoustic emission test will be done prior to therapy and q48 hours during their course of treatment with furosemide drip.

Dosage of furosemide drip, boluses and other relevant medications (i.e - vancomycin, muscular relaxants, aminoglycosides etc) will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* All children admitted to Pediatric ICU who are treated with furosemide continuous drip.

Exclusion Criteria:

* Children with known hearing abnormalities prior to treatment.

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: critically ill children in pediatric ICU.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2009-08; Study Completion 2010-08 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Elhanan Nahum, MD, Study Director — Schneider Children's Hospital
Locations (1):
- Pediatric ICU, Schneider Children's Hospital, Petah Tikva, Israel